CLINICAL TRIAL: NCT06920381
Title: Ethyl Chloride Spray to Reduce Pain From Local Anesthesia During Mohs Micrographic Surgery: A Randomized Clinical Trial
Brief Title: Ethyl Chloride Spray to Reduce Pain From Local Anesthesia During Mohs Micrographic Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2251013
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Surgery
Keywords: Mohs micrographic surgery; Ethyl Chloride Spray

STUDY DESIGN:
Intervention Model Description: This is a single-center, split-body study. The split-body design will involve dividing the surgical site into two equal halves, with one half (right side relative to patient) designated as the treatment side (receiving ethyl chloride spray prior to lidocaine injection) and the other as the control side (no ethyl chloride spray prior to injection).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ethyl Chloride Spray (Experimental): Prior to injection of lidocaine, the investigator will apply ethyl chloride spray, Gebauer's Ethyl Chloride Topical Spray, to the right side of the tumor lesion.
  This procedure will be performed for all patients participating in the trial.
  Interventions: Drug: Gebauer's Ethyl Chloride Topical Spray
- Control (No Intervention): The investigator will perform no intervention and will continue with the normal standard of care for injecting lidocaine into the left side of the tumor lesion.
  This procedure will be performed for all patients participating in the trial.

INTERVENTIONS:
Drug: Gebauer's Ethyl Chloride Topical Spray — Prior to injection of lidocaine, the investigator will apply ethyl chloride spray, Gebauer's Ethyl Chloride Topical Spray, continuously for 4 to 10 seconds until the skin turns white. This application will be done from a distance of 8 to 18 cm (3 to 7 inches) to the right side of the tumor lesion.
  Arms: Ethyl Chloride Spray

SUMMARY:
Fear of needles is a well-documented issue that affects many patients. This fear may cause significant anxiety in various medical situations, including in the dermatology office 1. If not properly managed, needle phobia can persist, affecting a patient's experience during each visit. This effect may compound and lead to avoidance behaviors that can delay necessary treatments 2. This issue is particularly relevant in a Mohs micrographic surgery (MMS) clinic where each patient experiences several painful needle injections before the day is over.

Ethyl chloride is gaining popularity among dermatologists for its routine use in clinical practice due to its anesthetic and antiseptic properties, especially as a pre-injection agent. Research indicates that cryotherapy or pre-cooling the skin before administering a local anesthetic may offer benefits over topical anesthetics, such as enhanced pain relief, quicker onset, and better patient compliance 3,4. However, to our knowledge, no studies have specifically examined the effectiveness of pre-cooling with ethyl chloride prior to Mohs micrographic surgery. To address this gap, we're conducting a trial aimed at evaluating the impact of pre-cooling with ethyl chloride on pain perception in adult patients undergoing Mohs micrographic surgery with local anesthetic injections.

The trial is a single-center, split-body study. The split-body design will involve dividing the surgical site into two equal halves, with one half (right side relative to patient) designated as the treatment side (receiving ethyl chloride spray prior to lidocaine injection) and the other as the control side (no ethyl chloride spray prior to injection). During the procedure, the participant will be asked to rate the pain associated with the needle injection AND the pain from infiltration of anesthetic from each side of the wound using the visual analog scale (VAS) scoring system (1 = no pain, 10 = most amount of pain possible). The results of the study will help us better understand how to mitigate pain and anxiety for patients requiring MMS.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for MMS with Dr. Daniel Eisen at UC Davis Health Department of Dermatology (3301 C St #1300-1400, Sacramento, CA 95816)
* Pre-op tumor size at least 1.5 cm (measured on day of procedure)

Exclusion Criteria:

* Skin disorders related to cold temperatures (i.e. cryoglobulinemia)
* Anxiolytic medication within past 4 hours
* Treatment sites around the eyes
* Pre-op tumor size smaller than 1.5 cm (measured on day of procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
VAS pain scores | During the MMS procedure
  The primary outcome measure will be the Visual Analog Scale (VAS) pain scores recorded at the time of the initial injection and during the infiltration of anesthetic for each treatment side. Patients will self-report their VAS score from a scale of 0-10. VAS scores will be sorted into 4 categories: 0 = no pain; 1-3 = mild pain; 4-6 = moderate pain; 7-10 = severe pain.
Subject response to "do you prefer precooling with ethyl chloride spray in future Mohs surgery cases?" | Immediately after the MMS procedure
  Secondary outcome measure will be study subject's responses to the question: "do you prefer precooling with ethyl chloride spray in future Mohs surgery cases?".

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Dermatology, Sacramento, California, United States

REFERENCES:
- [Result] Hamilton JG. Needle phobia: a neglected diagnosis. J Fam Pract. 1995 Aug;41(2):169-75. PMID 7636457
- [Result] Abbasi H, Ali F, Aslam H, Khan MS, Waqas M, Lal A. Cryoanesthesia with ethyl chloride spray versus 5% lidocaine gel in alleviating oral local anesthetic injection pain for buccal anaesthesia: A randomized clinical (controlled) trial. J Dent Res Dent Clin Dent Prospects. 2023 Winter;17(1):40-46. doi: 10.34172/joddd.2023.37041. Epub 2023 Apr 3. PMID 37650023
- [Result] Irkoren S, Ozkan HS, Karaca H. A Clinical Comparison of EMLA Cream and Ethyl Chloride Spray Application for Pain Relief of Forehead Botulinum Toxin Injection. Ann Plast Surg. 2015 Sep;75(3):272-4. doi: 10.1097/SAP.0000000000000121. PMID 25536197
- [Result] Flynn A, Barry R. Use of Ethyl Chloride in Dermatology Minor Surgery. Dermatol Surg. 2016 Mar;42(3):433-4. doi: 10.1097/DSS.0000000000000623. No abstract available. PMID 26849089
- [Result] Beroukhim K, Goldberg LH, Tarantino IS, Kimyai-Asadi A. The effect of intraoperative pain on patient satisfaction during Mohs micrographic surgery. J Am Acad Dermatol. 2022 Oct;87(4):848-849. doi: 10.1016/j.jaad.2021.10.025. Epub 2021 Oct 22. No abstract available. PMID 34695530
- [Result] Henke J, Immaneni S, Blalock T. Measuring pain and anxiety surrounding local anesthesia in Mohs micrographic surgery: A continuous and repeated-measure pilot study. J Am Acad Dermatol. 2023 Dec;89(6):1298-1300. doi: 10.1016/j.jaad.2023.08.039. Epub 2023 Aug 23. No abstract available. PMID 37625700
- [Result] Cooper DD, Seupaul RA. Does buffered lidocaine decrease the pain of local infiltration? Ann Emerg Med. 2012 Apr;59(4):281-2. doi: 10.1016/j.annemergmed.2011.05.025. Epub 2011 Aug 6. No abstract available. PMID 21820761
- [Result] Shilpapriya M, Jayanthi M, Reddy VN, Sakthivel R, Selvaraju G, Vijayakumar P. Effectiveness of new vibration delivery system on pain associated with injection of local anesthesia in children. J Indian Soc Pedod Prev Dent. 2015 Jul-Sep;33(3):173-6. doi: 10.4103/0970-4388.160343. PMID 26156269